CLINICAL TRIAL: NCT03388801
Title: Short and Long-term Follow-up of Quality-of-life and Pain After Spa Treatment in Elderly With Osteoarthritis
Brief Title: Quality-of-life and Pain After Spa Treatment in Elderly With Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Jolanta Zwolińska, Principal Investigator, University of Rzeszow
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Spa-osteoarthritis
Record Dates: First submitted 2017-12-01; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis; Quality of Life; Elderly; Balneology
MeSH Terms: conditions — Osteoarthritis | interventions — Balneology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spa therapy (Experimental): Spa treatment was applied during a session lasting 120 to 150 minutes a day. Spa treatment lasted 3 weeks, including treatments from Monday to Friday (15 days of treatment). As a part of comprehensive spa treatment, all the patients benefited from kinesiotherapy, physical agent modalities (electrotherapy, phototherapy), massage and balneotherapy (peloid therapy, hydrotherapy with mineral waters, crenotherapy).
  Interventions: Other: Spa therapy

INTERVENTIONS:
Other: Spa therapy — Spa treatment was applied during a session lasting 120 to 150 minutes a day. Spa treatment lasted 3 weeks, including treatments from Monday to Friday (15 days of treatment). As a part of comprehensive spa treatment, all the patients benefited from kinesiotherapy, physical agent modalities (electrotherapy, phototherapy), massage and balneotherapy (peloid therapy, hydrotherapy with mineral waters, crenotherapy).
  Other Names: balneotherapy

SUMMARY:
The aim of the study was to evaluate the short- and long-term effects of spa therapy on quality of life and pain in patients aged 65 years and older with osteoarthritis.

70 patients with osteoarthritis referred to spa treatment in south-eastern Poland were enrolled in the study. Spa treatment lasted 3 weeks.

All the patients benefited from spa therapy.

VAS pain scale, the Laitinen scale and WHOQOL-BREF questionnaire were used to assess the condition of the patients. The examinations were performed three times: at the beginning of the spa treatment, after three months and one year after the first examinations.

DETAILED DESCRIPTION:
In an interventional study design, there have been examined patients aged over 65 years with the diagnosis of osteoarthritis who were prescribed a first spa therapy course in spa resorts in south-eastern Poland, between April 2016 and July 2016.

Patients were assessed by an experienced physicians on the first day of the spa therapy (study 1), after three months (study 2) and one year (study 3) after the completion of the spa therapy.

All patients who had been enrolled to the study, were asked to fill out the appropriate questionnaires (on the first day of the spa therapy). The investigators ensured that questionnaires were properly completed, under the supervision of researcher previously trained for their application. Second (study 2) and third (study 3) stages of the study were performed after three months, and one year after the first study, respectively (participants were interviewed by telephone survey).

Interventions Spa treatment was applied during a session lasting 120 to 150 minutes a day. Spa treatment lasted 3 weeks, including treatments from Monday to Friday (15 days of treatment). As a part of comprehensive spa treatment, all the patients benefited from kinesiotherapy, physical agent modalities (electrotherapy, phototherapy), massage and balneotherapy (peloid therapy, hydrotherapy with mineral waters, crenotherapy).

ELIGIBILITY:
Inclusion Criteria:

* age over 65
* diagnosis of osteoarthritis,
* completion of 3 weeks of spa treatment
* patient's consent to participate in the study

Exclusion Criteria:

* failure to complete 3-weeks spa treatment,
* significant random events during follow-up
* diagnosed other diseases during follow-up,
* other forms of therapy implemented during follow-up,
* refusal to participate in II or III stage of the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Change in the quality of life | at baseline, 3 and 12 months
  Comparison of the WHOQOL-BREF questionnaire mean between baseline, 3 and 12 months. Quantitative evaluation of the primary outcome.

SECONDARY OUTCOMES:
Change in pain perception (VAS) | at baseline, 3 and 12 months
  Evolution of VAS (Visual Analogic Scale) between baseline, 3 and 12 months.
Change in: pain intensity, frequency of pain, frequency of using painkillers and mobility | at baseline, 3 and 12 months
  Evolution of the Modified Laitinen Pain Questionnaire between baseline, 3 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Zwolińska, Dr, Principal Investigator — Medical Faculty, University of Rzeszów

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zwolinska J, Weres A, Wyszynska J. One-Year Follow-Up of Spa Treatment in Older Patients with Osteoarthritis: A Prospective, Single Group Study. Biomed Res Int. 2018 Jul 2;2018:7492106. doi: 10.1155/2018/7492106. eCollection 2018. PMID 30065943